CLINICAL TRIAL: NCT02756754
Title: Radiofrequency Ablation for Aldosterone-producting Adenoma in Patients With Primary Aldosteronism: Evaluation of the Blood Pressure Control and of Its Safety.
Brief Title: Radiofrequency Ablation for Aldosterone-producting Adenoma in Patients With Primary Aldosteronism
Acronym: ADERADHTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15 7833 08
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Primary Aldosteronism; Adrenal Adenoma
MeSH Terms: conditions — Hyperaldosteronism; ACTH Syndrome, Ectopic | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiofrequency ablation (Experimental): Radiofrequency ablation (RFA) is a minimally invasive technique for eliminating both primary tumors and metastases.
  The needles that will be used are monopolar RFA, the LeVeen™ Needle Electrode Family with a generator "RF 3000" by Boston Scientific. The radiofrequency system will be used as the RFA generator device standard cycle of ablation will be applied in the patient. During RFA, blood pressure, pulse and oxygen saturation will be continuously monitored.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — The radiofrequency system will be used as the RFA generator device standard cycle of ablation will be applied in the patient. During RFA, blood pressure, pulse and oxygen saturation will be continuously monitored.

SUMMARY:
The aim of the study is to evaluate the novel use of adrenal radiofrequency ablation on a prospective cohort of patients with primary aldosteronism and unilateral adrenal adenoma concerning the efficacy on blood pressure control. The safety of the procedure is one of the secondary outcomes.

DETAILED DESCRIPTION:
The prevalence of hypertension dramatically increased. Although most cases of hypertension are idiopathic, some cases have an identifiable cause. Primary Aldosteronism (PA) is the most common cause of secondary hypertension and can be cured by surgery if PA is due to unilateral unique adrenal adenoma. Then this cause is worth identifying it. The surgery despite its minimally invasive nature is limited by the need for general anesthesia, the risk of vascular or visceral injuries, hematomas and all the adrenal gland is mostly removed. Imaged-guided percutaneous adrenal radiofrequency ablation (ARF) offers a less invasive alternative therapeutic option. This local therapy is employed to treat solid neoplasms whereas its application on functional adrenal adenoma is less documented and only a few case series with limited sample size are published. The impact on blood pressure control is not clearly reported. ARF ablation works by delivering a high-frequency alternating current through a needle electrode. An ionic agitation occurs and generates frictional heat for cell destruction at a predictable temperature and volume. Patients with a conventional documented PA due to unilateral adrenal nod who consented to the study were hospitalized. Patients with PA due to an aldosterone-producing adenoma are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* hypertension confirmed with ambulatory blood pressure monitoring
* primary aldosteronism demonstrated by hormonal assays: active renin (pg/ml) or plasma renin activity (ng/ml/h) and plasma aldosterone measured twice at baseline after an overnight fast, in sitting or recumbent position
* selective adrenal venous sampling after 40 years of age
* unilateral adrenal nod on CT scan <4cm
* adrenal radiofrequency ablation procedure of judged technically possible by radiologists

Exclusion Criteria:

* bilateral adrenal nods
* primary aldosteronism due to bilateral adrenal hyperplasia or macronodular hyperplasia
* lack of documented primary aldosteronism
* maximum tumor diameter greater than 4 cm
* Cushing syndrome or Pheochromocytoma
* when adrenal venous sampling is refused by the patient
* coagulopathy
* pregnant women
* patient with potentially inaccessible nodule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
mean day-time systolic/diastolic blood pressure | 6 months
  mean day-time systolic/diastolic blood pressure <135/85 mmHg at six months assessed by ambulatory blood pressure monitoring without antihypertensive treatment or a decrease of daytime systolic blood pressure of 20 mmHg and of diastolic blood pressure of 10 mmHg between baseline and 6 months

SECONDARY OUTCOMES:
day-time systolic and diastolic blood pressure | 6 months
  To assess a decrease of day-time systolic blood pressure of 20 mmHg and of diastolic blood pressure of 10 mmHg between baseline and 6 months
mean 24 hours systolic/diastolic blood pressure | 6 months
  mean 24 hours systolic/diastolic blood pressure <130/80 mmHg at six months assessed by ambulatory blood pressure monitoring without antihypertensive treatment
mean day-time ambulatory blood pressure | 6 months
  mean day-time ambulatory blood pressure changes assessed by ambulatory blood pressure monitoring between baseline and 6 months
mean night-time ambulatory blood pressure | 6 months
  mean night-time ambulatory blood pressure changes assessed by ambulatory blood pressure monitoring between baseline and 6 months
mean 24 hour ambulatory blood pressure changes assessed by ambulatory blood pressure | 6 months
  mean 24 hour ambulatory blood pressure changes assessed by ambulatory blood pressure monitoring between baseline and 6 months
casual systolic blood pressure / diastolic blood pressure | 6 months
  casual systolic blood pressure / diastolic blood pressure <140/90 mmHg after adrenal radiofrequency ablation, at six months without antihypertensive treatment
decrease of casual systolic blood pressure | 6 months
  decrease of casual systolic blood pressure of 20 mmHg and of casual diastolic blood pressure of 10 mmHg between baseline and 6 months
mean daytime ambulatory blood pressure changes assessed by self-measurement | 6 months
  mean daytime ambulatory blood pressure changes assessed by self-measurement of blood pressure monitoring between baseline and 6 months
antihypertensive agents | 6 months
  number of antihypertensive agents at 6 months after adrenal radiofrequency ablation
kalemia | 6 months
  evaluation of kalemia at month 1 and month 6
CT Scan | 6 months
  description of the CT scan aspect of the adrenal gland after adrenal radiofrequency ablation
post-operative complications | 6 months
  post-operative complications including retroperitoneal hematoma, pneumothorax, pain, infection
cost-effectiveness | 6 months
  cost-effectiveness radiofrequency ablation

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice DULY-BOUHANICK, Pr, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU Bordeaux, Bordeaux
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa N, Mounie M, Gombault-Datzenko E, Boulestreau R, Cremer A, Delchier MC, Gosse P, Lagarde S, Lepage B, Molinier L, Papadopoulos P, Trillaud H, Rousseau H, Bouhanick B. Cost Analysis of Radiofrequency Ablation for Adrenal Adenoma in Patients with Primary Aldosteronism and Hypertension: Results from the ADERADHTA Pilot Study and Comparison with Surgical Adrenalectomy. Cardiovasc Intervent Radiol. 2023 Jan;46(1):89-97. doi: 10.1007/s00270-022-03295-9. Epub 2022 Nov 15. PMID 36380152